CLINICAL TRIAL: NCT01574859
Title: Central Hypothyroidism and Cardiovascular Risk Factors
Brief Title: Central Hypothyroidism and Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ulla Feldt-Rasmussen, Professor, Rigshospitalet, Denmark
Other Study IDs: T4-CVR-12; T4-CVR-12 (Other Grant/Funding Number: Rigshospitalet)
Record Dates: First submitted 2012-04-07; First posted 2012-04-10 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Hypopituitarism
Keywords: central hypothyroidism; hypopituitarism; levothyroxine replacement; lipids; body composition
MeSH Terms: conditions — Hypopituitarism; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hypopituitarism: group of patients with hypopituitarism
  Interventions: Other: levothyroxine

INTERVENTIONS:
Other: levothyroxine — titration of T4 according to biochemical values

SUMMARY:
Retrospective trial of 300 patients with pituitary insufficiency treated in Department of Medica Endocrinology, Rigshospitalet, Copenhagen University concerning levothyroxine (T4) replacement and cardiovascular risk factors. The hypothesis is that subtle central hypothyroidism is associated with adverse cardiac risk factors, such as body composition and serum lipids, and that improved T4 replacement will eliminate this increased risk, independently of other pituitary hormone replacements.

DETAILED DESCRIPTION:
Retrospective trial of 300 patients with pituitary insufficiency treated in Department of Medical Endocrinology, Rigshospitalet, Copenhagen University concerning levothyroxine (T4) replacement and cardiovascular risk profile. The patient files are recruited among hypopituitary patients treated with growth hormone from the period 1993 to 2008. The trial is a retrospective assessment of data already collected for routine purposes and thus an audit of daily clinical practice. All information on the patients is obtained from the paper and electronic files existing in the department and no new measurements are foreseen.

ELIGIBILITY:
Inclusion Criteria:

* All patients with pituitary hypopituitarism

Exclusion Criteria:

* Unavailability of data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients at Rigshospitalet treated for pituitary hypothyroidism in the years 1993 to 2008
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
cholesterol | March 2002 - March 2013

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark